CLINICAL TRIAL: NCT00058448
Title: Phase II Study Of Weekly Docetaxel In Patients With Advanced Epidermoid Carcinoma Of The Penis
Brief Title: S0224, Docetaxel in Treating Patients With Locally Advanced or Metastatic Penile Cancer (TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to poor patient recruitment.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000297621; S0224 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2013-04

CONDITIONS: Penile Cancer
Keywords: stage II penile cancer; stage III penile cancer; stage IV penile cancer
MeSH Terms: conditions — Penile Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as docetaxel use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel in treating patients who have locally advanced or metastatic penile cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the confirmed complete and partial response rate in patients with locally advanced or metastatic epidermoid carcinoma of the penis treated with docetaxel.
* Determine the progression-free and overall survival of patients treated with this drug.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.

OUTLINE: Patients receive docetaxel IV over 15-30 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 3-5.8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed epidermoid carcinoma of the penis

  * Distant metastases (M1) OR
  * Pathologically confirmed regional nodal metastases (N1-3)
* Measurable disease

  * Soft tissue disease irradiated within the past 2 months is not considered measurable disease

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* White blood cell (WBC) count at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* Aspartate aminotransferase (SGOT) no greater than 2.5 times ULN

  * If SGOT is greater than ULN, alkaline phosphatase must be no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 4 times ULN

  * If alkaline phosphatase is greater than ULN, SGOT must be no greater than 1.5 times ULN

Renal

* Not specified

Other

* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II cancer currently in complete remission
* No grade 2 or greater peripheral neuropathy
* No hypersensitivity to drugs formulated with polysorbate 80 (e.g., recombinant interferon alfa-2a, multivitamin infusion, etoposide, infliximab, or NovoSeven factor)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for penile cancer

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 28 days since prior radiotherapy and recovered

Surgery

* Not specified

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria every 8 weeks during treatment | up to 24 weeks during treatment

SECONDARY OUTCOMES:
Safety as measured by Common Terminology Criteria for Adverse Events (CTC) Version 3.0 every 4 weeks | up to 24 weeks during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M. Beer, MD, Study Chair — OHSU Knight Cancer Institute; Roland T. Skeel, MD, Study Chair — Medical University of Ohio Cancer Center
Locations (49):
- United States (49):
  - St. Anthony Central Hospital, Denver, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - St. Anthony North Hospital, Westminster, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Salina Regional Health Center, Salina, Kansas
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Welch Cancer Center, Sheridan, Wyoming